CLINICAL TRIAL: NCT05588349
Title: Effectiveness of Trigger Point Dry Needling on Plantar Fasciitis: a Randomized Controlled Trial
Brief Title: Effectiveness of Trigger Point Dry Needling on Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Wing Sze, Student, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChineseUHK2022
Record Dates: First submitted 2022-10-15; First posted 2022-10-20 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Plantar Fascitis
Keywords: Plantar fasciitis; Dry needling
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Dry Needling; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Dry needling plus stretching exercise versus stretching exercise alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling + stretching exercise (Experimental): After locating the MTrPs, hand hygiene of the physiotherapist will be done and the needling site will be disinfected with alcohol swab. 0.30 x 50 mm disposable stainless-steel needles (DongBang Acupuncture Inc., Boryeong, Korea) will be used. The needle will be inserted into the muscle and pistoned in an up-and-down fashion using the "fast in and fast out" technique in order to provoke the local twitch response (LTR). This will be repeated until either the LTRs are exhausted, or the participant's tolerance threshold is met. If the participant is sensitive to the needle stimulation, the manipulation will be reduced. The needle will be left in situ for five minutes (Cotchett et al., 2011). Participants will receive dry needling once per week for three weeks. Plantar fascia and calf stretching exercise will be taught
  Interventions: Other: Dry needling
- Stretching exercise (Active Comparator): Plantar fascia stretching exercise:
  Participants will be instructed to sit with the affected foot placed on the contralateral thigh with the toes being grasped and pulled into extension until a stretch is felt in the plantar fascia.
  Calf stretching exercise:
  To focus on stretching the gastrocnemius, participants will be taught to stand with both hands holding onto the wall and keep the affected leg back with knee straightened and heel in contact with the floor. Slowly lean forward to the wall until a stretch is felt in the calf. To focus on stretching the soleus, the same procedures will be taught except with the affected knee being bent.
  Interventions: Other: Stretching exercise

INTERVENTIONS:
Other: Dry needling — Dry needling + stretching exercise
  Arms: Dry needling + stretching exercise
Other: Stretching exercise — Stretching exercise only
  Arms: Stretching exercise

SUMMARY:
Plantar fasciitis could lead to pain, disability and impaired balance. Dry needling that targets myofascial trigger points (MTrPs) has been shown to be beneficial in reducing pain, improving range of motion and function in patients with musculoskeletal conditions. Previous systematic review suggested a positive effect of dry needling on improving pain intensity and pain-related disability in patients with plantar heel pain (Llurda-Almuzara et al., 2021). However, the generalisability of the result is limited by small number of trials and heterogenicity in the dry needling application. Also, there is currently no evidence on its effect on dynamic balance and ankle dorsiflexion range of motion. This randomized controlled trial is designed to investigate the effectiveness of dry needling on pain, pain-related disability, dynamic balance and ankle dorsiflexion range of motion in patients with plantar fasciitis.

DETAILED DESCRIPTION:
Twenty participants aged 18 - 65 years with plantar fasciitis will be recruited and randomized to (1) dry needing and stretching exercise group or (2) stretching exercise group, receiving three treatment sessions over three weeks. The primary outcome measure will be numeric pain rating scale (NPRS) and the secondary outcome measures will be Chinese Foot and Ankle Outcome Score (FAOS), modified Star Excursion Balance Test (mSEBT) and weight bearing lunge test (WBLT) measured at baseline and week 4.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-65 years
* Clinical diagnosis of plantar fasciitis in accordance with the clinical guidelines of the Orthopaedic Section of the American Physical Therapy Association (APTA)
* Pain intensity of a minimum score of 5 on 11-point NPRS
* Presence of trigger points of the gastrocnemius or soleus muscles or both
* History of plantar heel pain for over 1 month

Exclusion Criteria:

* Needle allergy or phobia
* Bleeding disorders or severe vascular disease
* Pregnancy
* Cancer
* Fracture or surgery in the foot region or leg
* Infection
* Dermatological disease in the area of needling
* History of injection therapy in the heel during the previous three months
* Cognitive impairment
* Neurological disorders affecting balance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in first-step pain intensity | Baseline to 4 weeks
  The change in first-step pain intensity will be measured by the numeric pain rating scale (NPRS), which is a 11-point scale ranging from 0 ("no pain") to 10 ("the worst pain imaginable").

SECONDARY OUTCOMES:
Change in pain-related disability | Baseline to 4 weeks
  The change in pain-related disability will be measured by the Chinese Foot and Ankle Outcome Score (FAOS), which is a 42-item patient-reported outcome measure with a normalized score ranging from 0 to 100. A score of 100 resembling no symptoms and 0 resembling severe symptoms.
Change in dynamic balance | Baseline to 4 weeks
  The change in dynamic balance will be measured by the modified Star Excursion Balance Test (mSEBT). Participants stand on the leg to be tested and attempt to reach as far as possible with the reaching foot in 3 directions (anterior, posteromedial and posterolateral). The maximal distance reached along each direction (in centimeters) will be recorded. Greater reaching distance indicates better performance in dynamic balance.
Change in weight bearing ankle dorsiflexion range of motion | Baseline to 4 weeks
  The change in weight bearing ankle dorsiflexion range of motion will be measured by weight bearing lunge test (WBLT). Participants lunge forward until the knee could only make a slight contact with the wall with the heel remain in contact with the ground. The maximal distance (in centimeters) from the wall to the tip of the great toe is recorded. Greater distance indicates greater ankle dorsiflexion range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady of Maryknoll Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llurda-Almuzara L, Labata-Lezaun N, Meca-Rivera T, Navarro-Santana MJ, Cleland JA, Fernandez-de-Las-Penas C, Perez-Bellmunt A. Is Dry Needling Effective for the Management of Plantar Heel Pain or Plantar Fasciitis? An Updated Systematic Review and Meta-Analysis. Pain Med. 2021 Jul 25;22(7):1630-1641. doi: 10.1093/pm/pnab114. PMID 33760098
- [Background] Cotchett MP, Landorf KB, Munteanu SE, Raspovic AM. Consensus for dry needling for plantar heel pain (plantar fasciitis): a modified Delphi study. Acupunct Med. 2011 Sep;29(3):193-202. doi: 10.1136/aim.2010.003145. Epub 2011 Apr 18. PMID 21504939